CLINICAL TRIAL: NCT02369003
Title: Continuation of a Pilot Study to Evaluate the Safety and Feasibility of Implanting Autologous Peripheral Nerve Grafts in Subjects With Parkinson's Disease Undergoing Deep Brain Stimulation Surgery and Treatment
Brief Title: Cont. of a Study to Evaluate Implanting Peripheral Nerve Grafts Into Subjects With Parkinson's Disease (PD) During DBS
Acronym: CAPNG
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Craig van Horne, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Craig van Horne, MD, PhD, Principal Investigtator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-0729-F6A
Record Dates: First submitted 2015-01-12; First posted 2015-02-23 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; Schwann Cells
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peripheral Nerve Graft (Experimental): The intervention includes the surgical implantation of autologous peripheral nerve graft into the substantia nigra, basal forebrain, putamen, and/or STN of participants with Parkinson's Disease that are undergoing Deep Brain Stimulation (DBS).
  Interventions: Procedure: Autologous Peripheral Nerve Graft

INTERVENTIONS:
Procedure: Autologous Peripheral Nerve Graft — Implantation of Autologous Peripheral Nerve Graft into the substantia nigra, basal forebrain, putamen, and/or STN of participants with PD undergoing deep brain stimulation (DBS) surgery.

SUMMARY:
This pilot study is designed to follow up on a previous, preliminary study and test the long-term safety and feasibility of the implantation of autologous peripheral nerve grafts into the substantia nigra, basal forebrain, putamen, and/or STN of participants with PD undergoing deep brain stimulation (DBS) surgery. Peripheral nerve tissue contains Schwann cells which produce growth factors that have been demonstrated to support the survival and function of neurons.

Participants will serve as their own donor for the tissue, which will be implanted at the time they undergo DBS surgery.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to demonstrate safety of the approach: introducing a minor modification of a standard, FDA approved neurosurgical procedure in use for over a decade to implant autologous peripheral nerve into the central nervous system. As such, the study is designed to pose minimal risk and minimal inconvenience to the subjects. Additionally, the test paradigm is performed strategically to not interfere with the surgery or delivery of the scheduled clinical DBS therapy. The scientific basis for this study is that the implanted peripheral nerve tissue is naturally well suited to provide multiple growth factors that have been shown experimentally to support the survival and function of dopaminergic neurons. Central to this proposal is the hypothesis that the implanted tissue will physiologically deliver growth factors to restore to normal function the afflicted neurons found in PD.

The first specific aim is to assess the feasibility and safety of the combined peripheral nerve graft/DBS surgical procedure. The second specific aim is to evaluate the long term clinical safety of the peripheral nerve implant.

This pilot study will provide safety data that can be used to generate a larger phase III clinical trial. If successful, it would herald the development of a new treatment for PD in which patients are able to provide their own tissue as a source of growth factors that could arrest or reverse the ongoing cellular loss that is responsible for their devastating dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing DBS of the STN or GPi
* Between the ages of 40-75
* Able to give informed consent
* Show a positive response to Sinemet (carbidopa/levodopa)
* Be able to tolerate the surgical procedure

Exclusion Criteria:

* Any condition that would not make the subject a candidate for DBS of the STN or GPi
* Under the age of 40 or over the age of 75
* Unable to give informed consent
* Female who is pregnant, lactating, or of child-bearing potential unwilling to use an adequate birth control method during the period of the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 15 years
  Safety and Tolerability of Nerve Graft Implantation. Adverse events will be collected in order to measure the safety and tolerability of the grafting procedure. Adverse events will be documented and compared to the known and reported adverse events of DBS of Subthalamic Nucleus (STN) or internal globus pallidus (GPi).

SECONDARY OUTCOMES:
DaTscan assessment | 12 or 24 months
  Dopamine neurodegeneration at 12 or 24 months will be assessed using DaTscan SPECT imaging and compared to scans obtained before DBS surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Craig van Horne, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Background] Welleford AS, Quintero JE, Seblani NE, Blalock E, Gunewardena S, Shapiro SM, Riordan SM, Huettl P, Guduru Z, Stanford JA, van Horne CG, Gerhardt GA. RNA Sequencing of Human Peripheral Nerve in Response to Injury: Distinctive Analysis of the Nerve Repair Pathways. Cell Transplant. 2020 Jan-Dec;29:963689720926157. doi: 10.1177/0963689720926157. PMID 32425114
- [Background] van Horne CG, Quintero JE, Slevin JT, Anderson-Mooney A, Gurwell JA, Welleford AS, Lamm JR, Wagner RP, Gerhardt GA. Peripheral nerve grafts implanted into the substantia nigra in patients with Parkinson's disease during deep brain stimulation surgery: 1-year follow-up study of safety, feasibility, and clinical outcome. J Neurosurg. 2018 Dec 1;129(6):1550-1561. doi: 10.3171/2017.8.JNS163222. Epub 2018 Feb 18. PMID 29451447
- [Background] Aparicio GI, Quintero JE, Plum L, Deng L, Wanczyk K, Henry M, Lynch E, Murphy M, Gerhardt GA, van Horne CG, Monje PV. Identification of cellular and noncellular components of mature intact human peripheral nerve. J Peripher Nerv Syst. 2024 Sep;29(3):294-314. doi: 10.1111/jns.12643. Epub 2024 Jul 7. PMID 38973168
- [Background] Slevin JT, Gerhardt GA, Smith CD, Gash DM, Kryscio R, Young B. Improvement of bilateral motor functions in patients with Parkinson disease through the unilateral intraputaminal infusion of glial cell line-derived neurotrophic factor. J Neurosurg. 2005 Feb;102(2):216-22. doi: 10.3171/jns.2005.102.2.0216. PMID 15739547
- [Background] van Horne CG, Vaughan SW, Massari C, Bennett M, Asfahani WS, Quintero JE, Gerhardt GA. Streamlining deep brain stimulation surgery by reversing the staging order. J Neurosurg. 2015 May;122(5):1042-7. doi: 10.3171/2014.9.JNS14619. Epub 2015 Mar 6. PMID 25748305
- [Background] van Horne CG, Quintero JE, Gurwell JA, Wagner RP, Slevin JT, Gerhardt GA. Implantation of autologous peripheral nerve grafts into the substantia nigra of subjects with idiopathic Parkinson's disease treated with bilateral STN DBS: a report of safety and feasibility. J Neurosurg. 2017 Apr;126(4):1140-1147. doi: 10.3171/2016.2.JNS151988. Epub 2016 May 6. PMID 27153166
- [Background] Chau MJ, Quintero JE, Monje PV, Voss SR, Welleford AS, Gerhardt GA, van Horne CG. Using a Transection Paradigm to Enhance the Repair Mechanisms of an Investigational Human Cell Therapy. Cell Transplant. 2022 Jan-Dec;31:9636897221123515. doi: 10.1177/09636897221123515. PMID 36169034
- [Result] Quintero JE, Slevin JT, Gurwell JA, McLouth CJ, El Khouli R, Chau MJ, Guduru Z, Gerhardt GA, van Horne CG. Direct delivery of an investigational cell therapy in patients with Parkinson's disease: an interim analysis of feasibility and safety of an open-label study using DBS-Plus clinical trial design. BMJ Neurol Open. 2022 Jul 14;4(2):e000301. doi: 10.1136/bmjno-2022-000301. eCollection 2022. PMID 35949912
- [Result] Gera G, Guduru Z, Yamasaki T, Gurwell JA, Chau MJ, Krotinger A, Schmitt FA, Slevin JT, Gerhardt GA, van Horne C, Quintero JE. Gait and Balance Changes with Investigational Peripheral Nerve Cell Therapy during Deep Brain Stimulation in People with Parkinson's Disease. Brain Sci. 2021 Apr 15;11(4):500. doi: 10.3390/brainsci11040500. PMID 33921079
- [Result] Colvett I, Gilmore A, Guzman S, Ledreux A, Quintero JE, Ginjupally DR, Gurwell JA, Slevin JT, Guduru Z, Gerhardt GA, van Horne CG, Granholm AC. Recipient Reaction and Composition of Autologous Sural Nerve Tissue Grafts into the Human Brain. J Clin Med. 2023 Sep 22;12(19):6121. doi: 10.3390/jcm12196121. PMID 37834764
- [Result] Quintero JE, Chau MJ, Slevin JT, Koehl L, Gurwell JA, Wallace E, Kryscio RJ, El Khouli R, Anderson-Mooney AJ, Schmitt FA, Gerhardt GA, van Horne CG. Two-year feasibility and safety of open-label autologous peripheral nerve tissue implantation during deep brain stimulation in patients with Parkinson's disease. J Parkinsons Dis. 2025 Mar;15(2):397-408. doi: 10.1177/1877718X241312409. Epub 2025 Feb 25. PMID 40007169